CLINICAL TRIAL: NCT03385239
Title: A Randomized, Double-blind, Placebo-Controlled, Dose-Ranging Phase 2 Study of ISIS 678354 Administered Subcutaneously to Patients With Hypertriglyceridemia and Established Cardiovascular Disease (CVD) or at a High Risk for CVD
Brief Title: Study of ISIS 678354 (AKCEA-APOCIII-LRx) in Participants With Hypertriglyceridemia and Established Cardiovascular Disease (CVD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akcea Therapeutics (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 678354-CS2
Record Dates: First submitted 2017-12-01; First posted 2017-12-28 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Hypertriglyceridemia; Cardiovascular Diseases
Keywords: AKCEA-APOCIII-LRx; IONIS-APOCIII-LRx; Dyslipidemia; Metabolic Disease; Hyperlipidemia; Cardiac Disease; Lipid Metabolism Disorders; Triglycerides High; Vascular Diseases
MeSH Terms: conditions — Hypertriglyceridemia; Cardiovascular Diseases; Dyslipidemias; Metabolic Diseases; Hyperlipidemias; Heart Diseases; Lipid Metabolism Disorders; Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Pooled Placebo (Placebo Comparator): Participants in each cohort (A, B, C and D) were randomized to receive placebo at a dose-matched volume of study drug (ISIS 678354).
  Interventions: Drug: Placebo
- Cohort A: ISIS 678354: 10 mg Q4W (Experimental): Cohort A participants received 10 milligrams (mg) ISIS 678354, subcutaneous (SC) injection, once every 4 weeks (Q4W), for up to 49 weeks and a maximum of 13 doses.
  Interventions: Drug: ISIS 678354
- Cohort C: ISIS 678354: 15 mg Q2W (Experimental): Cohort C participants received 15 mg ISIS 678354, SC injection, once every 2 weeks (Q2W) for up to 51 weeks and a maximum of 26 doses.
  Interventions: Drug: ISIS 678354
- Cohort D: ISIS 678354: 10 mg QW (Experimental): Cohort D participants received 10 mg ISIS 678354, SC injection, once weekly (QW) for up to 52 weeks and a maximum of 52 doses.
  Interventions: Drug: ISIS 678354
- Cohort B: ISIS 678354: 50 mg Q4W (Placebo Comparator): Cohort B participants received 50 mg ISIS 678354, SC injection, once Q4W for up to 49 weeks and a maximum of 13 doses.
  Interventions: Drug: ISIS 678354

INTERVENTIONS:
Drug: ISIS 678354 — ISIS 678354 solution for SC injection.
  Other Names: AKCEA-APOCIII-LRx, IONIS-APOCIII-LRx
  Arms: Cohort A: ISIS 678354: 10 mg Q4W; Cohort B: ISIS 678354: 50 mg Q4W; Cohort C: ISIS 678354: 15 mg Q2W; Cohort D: ISIS 678354: 10 mg QW
Drug: Placebo — Sterile Normal Saline (0.9% NaCl).
  Arms: Pooled Placebo

SUMMARY:
This was a multicenter, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the safety, including tolerability, of ISIS 678354 and to assess the efficacy of different doses and dosing regimens of ISIS 678354 for reduction of serum triglyceride (TG) levels in participants with hypertriglyceridemia and established CVD or at a high risk for CVD.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of CVD (defined as documented coronary artery disease, stroke, or peripheral artery disease).
* Fasting serum triglycerides (TG) greater than or equal to (≥) 200 milligrams per deciliter (mg/dL) (≥ 2.3 millimoles per liter (mmol/L)) and less than or equal to (≤) 500 mg/dL (≥ 5.7 mmol/L) at Screening.
* Fasting TG ≥ 200 mg/dL and ≤ 500 mg/dL at Qualification visit.
* Must be on standard-of-care preventative therapy for known CVD risk factors.

Key Exclusion Criteria:

* Within 6 months of Screening: acute coronary syndrome, major cardiac surgery, or stroke/transient ischemic attack (TIA).
* Within 3 months of Screening: coronary, carotid, or peripheral arterial revascularization, major non-cardiac surgery, or lipoprotein apheresis.
* Heart failure New York Heart Association (NYHA) class IV.
* Type 1 diabetes mellitus.
* Type 2 diabetes mellitus with any of the following:

  * Newly diagnosed within 12 weeks of Screening.
  * Glycated hemoglobin (HbA1c) ≥ 9.0% at Screening.
  * Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of Screening [with the exception of ± 10 units of insulin].
* Body Mass Index (BMI) greater than (>) 40 kilograms per square meter (kg/m^2).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (24):
  - Clinical Site, Cottonwood, Arizona
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Carmichael, California
  - Clinical Site, Fresno, California
  - Clinical Site, La Jolla, California
  - Clinical Site, Long Beach, California
  - Clinical Site, Montclair, California
  - Clinical Site, Wilmington, Delaware
  - Clinical Site, Boca Raton, Florida
  - Clinical Site, Jacksonville, Florida
  - Clinical Site, New Port Richey, Florida
  - Clinical Site, Munster, Indiana
  - Clinical Site, Ames, Iowa
  - Clinical Site, Kansas City, Kansas
  - Clinical Site, Louisville, Kentucky
  - Clinical Site, Fall River, Massachusetts
  - Clinical Site, Cooperstown, New York
  - Clinical Site, High Point, North Carolina
  - Clinical Site, Portland, Oregon
  - Clinical Site, Lansdale, Pennsylvania
  - Clinical Site, Providence, Rhode Island
  - Clinical Site, Greer, South Carolina
  - Clinical Site, Houston, Texas
  - Clinical Site, Milwaukee, Wisconsin
- Canada (7):
  - Clinical Site, Cambridge, Ontario
  - Clinical Site, Greater Sudbury, Ontario
  - Clinical Site, Brossard, Quebec
  - Clinical Site, Chicoutimi, Quebec
  - Clinical Site, Gatineau, Quebec
  - Clinical Site, Montreal, Quebec
  - Clinical Site, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tardif JC, Karwatowska-Prokopczuk E, Amour ES, Ballantyne CM, Shapiro MD, Moriarty PM, Baum SJ, Hurh E, Bartlett VJ, Kingsbury J, Figueroa AL, Alexander VJ, Tami J, Witztum JL, Geary RS, O'Dea LSL, Tsimikas S, Gaudet D. Apolipoprotein C-III reduction in subjects with moderate hypertriglyceridaemia and at high cardiovascular risk. Eur Heart J. 2022 Apr 6;43(14):1401-1412. doi: 10.1093/eurheartj/ehab820. PMID 35025993

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a clinical diagnosis of hypertriglyceridemia and established cardiovascular disease (CVD) or at high risk for CVD were enrolled in 32 study sites in United States and Canada between 30 January 2018 to 25 February 2020.
Pre-assignment Details: 114 participants were randomized in a 1:1:1:1 ratio to Cohorts A, B, C or D. In each cohort, participants were randomized in a 4:1 ratio to receive ISIS 678354 or placebo. Placebo participants from all cohorts were pooled for analysis and presented as the pooled placebo group.
Groups:
- Pooled Placebo: Participants in each cohort were randomized to receive placebo at a dose-matched volume of study drug (ISIS 678354).
Period: Overall Study
Arm/Group | Pooled Placebo | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
Started | 24 | 22 | 23 | 23 | 22
Completed (Completed here refers to participants who completed post-treatment follow-up.) | 22 | 19 | 20 | 19 | 22
Not Completed | 2 | 3 | 3 | 4 | 0
Not completed — Voluntary Withdrawal | 2 | 3 | 2 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized and received at least 1 dose of study drug (ISIS 678354 or placebo).
Groups:
- Cohort A: ISIS 678354: 10 mg Q4W: Cohort A participants received 10 mg ISIS 678354, SC injection, Q4W, for up to 49 weeks and a maximum of 13 doses.
- Cohort C: ISIS 678354: 15 mg Q2W: Cohort C participants received 15 mg ISIS 678354, SC injection, Q2W for up to 51 weeks and a maximum of 26 doses.
- Cohort D: ISIS 678354: 10 mg QW: Cohort D participants received 10 mg ISIS 678354, SC injection, QW for up to 52 weeks and a maximum of 52 doses.
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W | Total
Number analyzed (Participants) | 24 | 22 | 23 | 23 | 22 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (7.93) | 64.4 (9.13) | 68.9 (6.82) | 65.6 (8.48) | 62.9 (7.40) | 65.3 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 4 | 5 | 7 | 28
  Male | 20 | 14 | 19 | 18 | 15 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 1 | 0 | 7
  Not Hispanic or Latino | 23 | 19 | 21 | 22 | 22 | 107
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2 | 4
  White | 22 | 20 | 23 | 23 | 18 | 106
  More than one race | 0 | 1 | 0 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Fasting Triglycerides (TG) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 293.8 (86.68) | 281.6 (73.43) | 284.8 (94.54) | 292.3 (89.29) | 268.4 (85.08) | 284.4 (85.16)
Apolipoprotein CIII (ApoC-III) [Mean (Standard Deviation); unit: mg/dL] | 16.618 (4.4720) | 16.030 (4.1482) | 15.849 (4.2456) | 16.810 (4.2021) | 15.669 (3.2484) | 16.205 (4.0466)
Total Cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 144.8 (26.00) | 149.2 (28.81) | 163.1 (35.09) | 160.0 (34.55) | 166.8 (35.30) | 156.7 (32.66)
LDL Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 55.9 (26.06) | 62.4 (22.57) | 73.1 (29.73) | 71.2 (30.24) | 74.8 (22.47) | 67.4 (27.02)
HDL Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 34.6 (8.61) | 34.1 (9.07) | 33.9 (9.48) | 34.8 (8.61) | 36.8 (10.54) | 34.8 (9.16)
Non-HDL Cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 110.3 (23.96) | 115.1 (28.93) | 129.2 (33.32) | 125.3 (32.09) | 130.1 (31.02) | 121.9 (30.52)
VLDL Cholesterol (VLDL-C) [Mean (Standard Deviation); unit: mg/dL] | 54.9 (12.71) | 54.0 (10.99) | 56.1 (21.45) | 54.1 (11.80) | 55.2 (26.84) | 54.9 (17.51)
Apolipoprotein B (ApoB) [Mean (Standard Deviation); unit: mg/dL] | 77.1 (19.71) | 79.6 (16.55) | 87.9 (20.60) | 86.8 (19.62) | 88.5 (14.29) | 83.9 (18.65)
Apolipoprotein A1 (ApoA-I) [Mean (Standard Deviation); unit: mg/dL] | 131.4 (19.28) | 130.2 (19.15) | 129.0 (16.69) | 132.5 (22.95) | 136.3 (23.07) | 131.9 (20.14)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG) at the Primary Analysis Time Point
Description: An analysis of covariance (ANCOVA) model was performed on the log ratio of TG value at the Primary Analysis Time Point to TG value at Baseline. The estimate of the log ratio was converted back to the original scale and percent change was calculated using formula: (ratio of TG value at the Primary Analysis Time Point to TG value at Baseline - 1) × 100.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A and B and Week 27 for Cohorts C and D)
Population: FAS included all participants who were randomized and received at least 1 dose of study drug (ISIS 678354 or placebo). Here, 'Number analyzed' ('n') = Participants evaluable for this outcome measure at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Pooled Placebo | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
Number analyzed (Participants) | 24 | 22 | 23 | 23 | 22
percent change | 6 [-9 to 23] | -23 [-34 to -10] | -56 [-62 to -49] | -60 [-66 to -54] | -60 [-65 to -53]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; Test type: Superiority; p = 0.0042, ANCOVA; Mean Difference in % CFB = -27, 95% CI 2-sided [-41 to -10] — Mean difference in percent (%) change from baseline (CFB) based on difference in least square mean (LSM) of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -58, 95% CI 2-sided [-66 to -48] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -63, 95% CI 2-sided [-70 to -54] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -62, 95% CI 2-sided [-69 to -53] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE was considered to be related to the investigational drug product. A TEAE was defined as any AE starting on or after the first dose of the study drug.
Time Frame: Up to the 13-week post-treatment follow-up period (Up to approximately 15 months)
Population: Safety set included all participants who were randomized and received at least 1 dose of study drug (ISIS 678354 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
Number analyzed (Participants) | 24 | 22 | 23 | 23 | 22
Participants | 20 | 17 | 20 | 22 | 21

3. Secondary Outcome: Percent Change From Baseline in ApoC-III, TC, LDL-C, HDL-C, Non-HDL-C, VLDL-C, ApoB, and ApoA-I at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the log ratio of Primary Analysis Time Point value to Baseline value for ApoC-III, TC, LDL-C, HDL-C, Non-HDL-C, VLDL-C, ApoB, and ApoA-I. The estimate of the log ratio was converted back to the original scale and percent change for each lipid parameter was calculated using formula: (ratio of Primary Analysis Time Point value to Baseline value - 1) × 100.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A and B and Week 27 for Cohorts C and D)
Population: FAS included all participants who were randomized and received at least 1 dose of study drug (ISIS 678354 or placebo). Here, 'Number analyzed' ('n') = Participants evaluable for this outcome measure for each specified category.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Pooled Placebo | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
Number analyzed (Participants) | 24 | 22 | 23 | 23 | 22
percent change
  Apo-C III: number analyzed (Participants) | 20 | 18 | 18 | 18 | 21
  Apo-C III | 2 [-16 to 23] | -29 [-42 to -13] | -68 [-74 to -61] | -73 [-78 to -67] | -74 [-78 to -69]
  TC: number analyzed (Participants) | 20 | 18 | 19 | 18 | 21
  TC | 1 [-6 to 7] | -2 [-8 to 5] | -12 [-17 to -5] | -3 [-9 to 4] | -8 [-13 to -2]
  LDL-C: number analyzed (Participants) | 20 | 18 | 19 | 18 | 20
  LDL-C | -2 [-13 to 11] | 5 [-7 to 19] | 2 [-10 to 15] | 27 [13 to 44] | 10 [-2 to 23]
  HDL-C: number analyzed (Participants) | 20 | 18 | 19 | 18 | 21
  HDL-C | -1 [-8 to 6] | 11 [3 to 19] | 33 [24 to 43] | 40 [30 to 51] | 29 [20 to 39]
  Non-HDL-C: number analyzed (Participants) | 20 | 18 | 19 | 18 | 21
  Non-HDL-C | 1 [-8 to 10] | -6 [-15 to 3] | -24 [-31 to -17] | -15 [-23 to -7] | -19 [-26 to -12]
  VLDL-C: number analyzed (Participants) | 20 | 18 | 19 | 18 | 20
  VLDL-C | -2 [-13 to 11] | -22 [-32 to -12] | -54 [-59 to -48] | -59 [-63 to -53] | -60 [-65 to -55]
  ApoB: number analyzed (Participants) | 20 | 18 | 19 | 18 | 21
  ApoB | -2 [-8 to 5] | 0 [-7 to 8] | -17 [-23 to -12] | -7 [-13 to 0] | -12 [-18 to -6]
  ApoA-1: number analyzed (Participants) | 20 | 18 | 19 | 18 | 21
  ApoA-1 | 0 [-4 to 4] | 5 [1 to 10] | 14 [9 to 19] | 18 [13 to 23] | 14 [9 to 18]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; ApoC III; Test type: Superiority; p = 0.0123, ANCOVA; Mean Difference in % CFB = -30, 95% CI 2-sided [-47 to -8] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; Apo-C III; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -68, 95% CI 2-sided [-76 to -58] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; Apo-C III; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -74, 95% CI 2-sided [-80 to -65] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; Apo-C III; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -74, 95% CI 2-sided [-80 to -66] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 5: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; TC; Test type: Superiority; p = 0.568, ANCOVA; Mean Difference in % CFB = -3, 95% CI 2-sided [-11 to 7] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 6: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; TC; Test type: Superiority; p = 0.008, ANCOVA; Mean Difference in % CFB = -12, 95% CI 2-sided [-19 to -3] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 7: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; TC; Test type: Superiority; p = 0.4476, ANCOVA; Mean Difference in % CFB = -3, 95% CI 2-sided [-12 to 6] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 8: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; TC; Test type: Superiority; p = 0.0606, ANCOVA; Mean Difference in % CFB = -8, 95% CI 2-sided [-16 to 0] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 9: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; LDL-C; Test type: Superiority; p = 0.4509, ANCOVA; Mean Difference in % CFB = 7, 95% CI 2-sided [-10 to 26] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 10: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; LDL-C; Test type: Superiority; p = 0.6746, ANCOVA; Mean Difference in % CFB = 4, 95% CI 2-sided [-12 to 23] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 11: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; LDL-C; Test type: Superiority; p = 0.0032, ANCOVA; Mean Difference in % CFB = 29, 95% CI 2-sided [9 to 53] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 12: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; LDL-C; Test type: Superiority; p = 0.1996, ANCOVA; Mean Difference in % CFB = 12, 95% CI 2-sided [-6 to 32] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 13: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; HDL-C; Test type: Superiority; p = 0.0373, ANCOVA; Mean Difference in % CFB = 12, 95% CI 2-sided [1 to 24] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 14: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; HDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = 34, 95% CI 2-sided [21 to 49] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 15: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; HDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = 42, 95% CI 2-sided [28 to 57] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 16: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; HDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = 30, 95% CI 2-sided [18 to 44] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 17: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; Non-HDL-C; Test type: Superiority; p = 0.2826, ANCOVA; Mean Difference in % CFB = -7, 95% CI 2-sided [-18 to 6] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 18: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; Non-HDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -24, 95% CI 2-sided [-34 to -14] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 19: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; Non-HDL-C; Test type: Superiority; p = 0.0118, ANCOVA; Mean Difference in % CFB = -15, 95% CI 2-sided [-26 to -4] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 20: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; Non-HDL-C; Test type: Superiority; p = 0.0009, ANCOVA; Mean Difference in % CFB = -20, 95% CI 2-sided [-29 to -9] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 21: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; VLDL-C; Test type: Superiority; p = 0.0086, ANCOVA; Mean Difference in % CFB = -21, 95% CI 2-sided [-34 to -6] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 22: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; VLDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -53, 95% CI 2-sided [-60 to -44] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 23: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; VLDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -58, 95% CI 2-sided [-64 to -50] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 24: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; VLDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -60, 95% CI 2-sided [-66 to -52] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 25: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; ApoB; Test type: Superiority; p = 0.6801, ANCOVA; Mean Difference in % CFB = 2, 95% CI 2-sided [-7 to 13] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 26: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; ApoB; Test type: Superiority; p = 0.0007, ANCOVA; Mean Difference in % CFB = -16, 95% CI 2-sided [-24 to -7] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 27: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; ApoB; Test type: Superiority; p = 0.3183, ANCOVA; Mean Difference in % CFB = -5, 95% CI 2-sided [-14 to 5] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 28: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; ApoB; Test type: Superiority; p = 0.024, ANCOVA; Mean Difference in % CFB = -10, 95% CI 2-sided [-19 to -1] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 29: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; ApoA-I; Test type: Superiority; p = 0.0936, ANCOVA; Mean Difference in % CFB = 5, 95% CI 2-sided [-1 to 11] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 30: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; ApoA-I; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = 14, 95% CI 2-sided [8 to 21] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 31: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; ApoA-I; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = 18, 95% CI 2-sided [11 to 25] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 32: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; ApoA-I; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = 14, 95% CI 2-sided [7 to 20] — Mean difference in % CFB based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated

4. Secondary Outcome: Percentage of Participants Who Achieved Fasting Triglycerides (TG) <= 150 mg/dL (<= 1.7 Millimoles Per Liter [mmol/L])
Description: The percentage of participants who achieved <= 150 mg/dL or <= 1.7 mmol/L of fasting TG levels at the primary analysis time point were compared between each ISIS 678354 treatment group and pooled placebo group using a logistic regression model with log-transformed baseline TG value as a covariate.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A and B and Week 27 for Cohorts C and D)
Population: FAS included all participants who were randomized and received at least 1 dose of study drug (ISIS 678354 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
Number analyzed (Participants) | 24 | 22 | 23 | 23 | 22
percentage of participants | 4.2 | 13.6 | 65.2 | 73.9 | 90.9
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; Test type: Superiority; p = 0.2591, Regression, Logistic; Odds Ratio (OR) = 3.34, 95% CI 2-sided [0.41 to 27.20]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 84.02, 95% CI 2-sided [9.54 to 740.02]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 322.79, 95% CI 2-sided [20.31 to 5130.99]
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 342.13, 95% CI 2-sided [23.72 to 4933.89]

5. Secondary Outcome: Percentage of Participants Who Achieved Fasting Triglycerides (TG) <= 100 mg/dL (<= 1.13 mmol/L)
Description: The percentage of participants who achieved <= 100 mg/dL or <= 1.13 mmol/L of fasting TG levels at the primary analysis time point were compared between each ISIS 678354 treatment group and pooled placebo group using a logistic regression model with log-transformed baseline TG value as a covariate.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A and B and Week 27 for Cohorts C and D)
Population: FAS included all participants who were randomized and received at least 1 dose of study drug (ISIS 678354 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
Number analyzed (Participants) | 24 | 22 | 23 | 23 | 22
percentage of participants | 0 | 0 | 30.4 | 26.1 | 45.5
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: ISIS 678354: 10 mg Q4W; Test type: Superiority; p = 0.9119, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.02 to 69.88]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 678354: 15 mg Q2W; Test type: Superiority; p = 0.0306, Regression, Logistic; Odds Ratio (OR) = 27.18, 95% CI 2-sided [1.36 to 542.48]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort D: ISIS 678354: 10 mg QW; Test type: Superiority; p = 0.0344, Regression, Logistic; Odds Ratio (OR) = 25.54, 95% CI 2-sided [1.27 to 514.20]
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 678354: 50 mg Q4W; Test type: Superiority; p = 0.0123, Regression, Logistic; Odds Ratio (OR) = 44.47, 95% CI 2-sided [2.28 to 866.49]

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of ISIS 678354
Time Frame: Predose, 1, 2, 4, 8, 24 hours post the first dose (Day 1), Week 21 (for Cohorts A and B) and Week 25 (for Cohorts C and D)
Population: Pharmacokinetic (PK) subgroup: Subset of participants who were randomized, received at least (>=) 1 dose of ISIS 678354, had >= 1 evaluable concentration result post first dose and had additional PK sampling after dose administration on Day 1 and Week 21 (Cohorts A and B) or Week 25 (Cohorts C and D). 'Number analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
Number analyzed (Participants) | 5 | 8 | 4 | 2
nanograms per milliliter (ng/mL)
  Day 1 | 53.7 (181.2) | 45.9 (36.2) | 35.8 (71.1) | 48.8 (333.3)
  Week 21 (for Cohorts A and B) and Week 25 (for Cohorts C and D): number analyzed (Participants) | 5 | 7 | 2 | 2
  Week 21 (for Cohorts A and B) and Week 25 (for Cohorts C and D) | 41.0 (324.1) | 48.0 (29.9) | 45.1 (47.4) | 127 (29.9)

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of ISIS 678354
Time Frame: as for outcome 6
Population: PK subgroup: Subset of participants who were randomized, received >= 1 dose of ISIS 678354, had >= 1 evaluable concentration result post first dose and had additional PK sampling after dose administration on Day 1 and Week 21 (Cohorts A and B) or Week 25 (Cohorts C and D). 'Number analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
Number analyzed (Participants) | 5 | 8 | 4 | 2
hours (h)
  Day 1 | 1.08 [1.00 to 2.00] | 2.00 [1.98 to 4.00] | 3.03 [2.00 to 4.00] | 1.50 [1.05 to 1.95]
  Week 21 (for Cohorts A and B) and Week 25 (for Cohorts C and D): number analyzed (Participants) | 5 | 7 | 2 | 2
  Week 21 (for Cohorts A and B) and Week 25 (for Cohorts C and D) | 2.00 [0.917 to 8.00] | 2.08 [1.00 to 4.00] | 2.50 [1.00 to 4.00] | 4.04 [4.02 to 4.07]

8. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours (AUC0-24) of ISIS 678354
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
Number analyzed (Participants) | 5 | 8 | 4 | 2
nanograms*hours per milliliter (ng*h/mL)
  Day 1 | 618 (115.6) | 499 (31.1) | 411 (59.0) | 563 (334.6)
  Week 21 (for Cohorts A and B) and Week 25 (for Cohorts C and D): number analyzed (Participants) | 5 | 7 | 2 | 2
  Week 21 (for Cohorts A and B) and Week 25 (for Cohorts C and D) | 468 (258.4) | 499 (11.2) | 454 (26.3) | 1460 (13.6)

ADVERSE EVENTS:
Time Frame: Up to the 13-week post-treatment follow-up period (Up to approximately 15 months)
Description: Safety set included all participants who were randomized and received at least 1 dose of study drug (ISIS 678354 or placebo).
Arm/Group | Pooled Placebo | Cohort A: ISIS 678354: 10 mg Q4W | Cohort C: ISIS 678354: 15 mg Q2W | Cohort D: ISIS 678354: 10 mg QW | Cohort B: ISIS 678354: 50 mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22 | 1/23 | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/24 | 3/22 | 4/23 | 1/23 | 3/22
Other Adverse Events (participants affected / at risk) | 16/24 | 15/22 | 19/23 | 20/23 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=24) | Cohort A: ISIS 678354: 10 mg Q4W (N=22) | Cohort C: ISIS 678354: 15 mg Q2W (N=23) | Cohort D: ISIS 678354: 10 mg QW (N=23) | Cohort B: ISIS 678354: 50 mg Q4W (N=22)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Post polio syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=24) | Cohort A: ISIS 678354: 10 mg Q4W (N=22) | Cohort C: ISIS 678354: 15 mg Q2W (N=23) | Cohort D: ISIS 678354: 10 mg QW (N=23) | Cohort B: ISIS 678354: 50 mg Q4W (N=22)
Nasopharyngitis (Infections and infestations) | 3 | 3 | 4 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 3 | 4 | 3
Urinary tract infection (Infections and infestations) | 1 | 2 | 2 | 1 | 4
Bronchitis (Infections and infestations) | 2 | 1 | 2 | 2 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 2 | 0 | 3
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 2 | 3 | 5 | 4
Fatigue (General disorders) | 1 | 2 | 1 | 2 | 1
Non-cardiac chest pain (General disorders) | 2 | 2 | 2 | 0 | 1
Injection site pruritus (General disorders) | 0 | 1 | 1 | 2 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 2 | 1
Injection site haemorrhage (General disorders) | 1 | 1 | 0 | 2 | 0
Injection site pain (General disorders) | 0 | 2 | 0 | 1 | 0
Influenza like illness (General disorders) | 2 | 0 | 0 | 1 | 0
Pain (General disorders) | 2 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 3 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 2 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 2 | 3
Hypotension (Vascular disorders) | 1 | 2 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 2 | 1 | 0 | 2 | 1
Haemoglobin decreased (Investigations) | 2 | 0 | 1 | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 2 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 2 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT03385239/Prot_SAP_001.pdf